CLINICAL TRIAL: NCT00708604
Title: Islet After Kidney Transplantation (IAK) in Patients With Type 1 Diabetes Using a Sirolimus/Tacrolimus/MMF-Based Immunosuppressive Regimen
Brief Title: Islet After Kidney Transplantation (IAK) in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04033; DK56952
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Kidney Transplantation; Islet Transplantation; Sirolimus/Tacrolimus/MMF-based Immunosuppressive Regimen
MeSH Terms: conditions — Diabetes Mellitus | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Islet transplantation
  Interventions: Procedure: Islet Transplantation; Biological: Islet cell transplantation

INTERVENTIONS:
Procedure: Islet Transplantation — Islet Transplantation
Biological: Islet cell transplantation — Islet cell transplantation will occur through the portal vein.

SUMMARY:
The purpose of this study is to determine the safety of islet transplantation in patients with type 1 diabetes who have had a successful kidney transplant and have been maintained for at least three months on anti-rejection medications consisting of any combination of sirolimus, tacrolimus, MMF or prednisone (5 mg/day or less). Another purpose is to determine the effectiveness of an islet transplant in inducing insulin independence and whether or not an islet transplant improves quality of life for kidney transplants patients with type 1 diabetes.

DETAILED DESCRIPTION:
Insulin is a hormone that helps the body use sugar and keeps blood sugar levels normal. Special cells in the human body, called beta cells, make insulin. Beta cells are found inside small groups of cells called "islets." Islets are found scattered in the pancreas gland. Type 1 diabetes is caused by damage to these insulin-making cells. Type 1 diabetic patients need insulin shots because their body does not make enough insulin. Even with insulin shots, many diabetic patients develop damage to the heart, blood vessels, nerves, eyes and kidneys. Research studies suggest that these problems are caused by blood sugar levels being too high.

Another way to treat diabetes is by giving the patient a pancreas transplant. The pancreas transplant gives the patient new insulin-making cells. If the pancreas transplant works, the patient does not need insulin shots. Pancreas transplantation is considered major surgery, and things can go wrong after surgery. Transplantation of just the islets, and not the rest of the pancreas, can be done without a major surgery. Research doctors have been studying islet transplantation to determine whether subjects who undergo the procedure can get off insulin shots, without the dangers of a major surgery.

In 2000, a group of research doctors in Edmonton, Canada reported that 3 out of 4 research subjects given islet transplants from brain-dead donors did not need insulin shots for approximately 2 years after transplantation. The research doctors from Edmonton have also reported that most islet transplant recipients in their study start to need insulin shots again with longer follow-up. So far, only about 1 out of 10 of the research subjects in the original Edmonton trial remain off of insulin 5 years after their transplant. The reasons that islet transplants stop working well enough and the recipients need to start insulin again are not known at this time. As with any type of transplant, all of the research subjects receiving islets from donors needed medicine to stop their bodies from rejecting the transplants. This study uses a few additional medications/vitamins that were not included in the Edmonton study that may improve the long-term outcome of islet transplantation. Some research studies suggest that for subjects with type 1 diabetes, an islet transplant may also help the kidney transplant work better and last longer.

This study is being performed to confirm that islet after kidney transplantation (IAK) is a safe and effective procedure for kidney transplant patients with type 1 diabetes who are on any combination of sirolimus, tacrolimus, MMF or prednisone (5 mg per day or less) anti-rejection medications for the care of their kidney transplant. Subjects will be followed closely for two years after islet transplant to monitor blood sugar control, the health of the kidney transplant, and changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus. Documentation of negative basal and stimulated C-peptide (a basal level of </= 0.2 ng/ml before IV administration of 1 mg of glucagon, and a glucagon stimulated C-peptide </= 0.8 ng/ml) and diagnosis of diabetes for at least 5 years.
* Recipient of renal transplant with good function (serum creatinine </= 1.6 mg/dl, creatinine clearance >/=60 ml/min and albumin excretion </= 300 mg/24 hr) for >3 months.
* Stable immunosuppression consisting of any combination of sirolimus, tacrolimus, MMF or </= 5 mg/day of corticosteroids for at least 3 months, without major complications.
* No history of acute rejection episodes related to renal graft in last 12 months and low risk for developing acute rejection (first renal transplant, PRA <25%, negative kidney crossmatch by B, T, flow cytometry)
* Under the continuing care of a renal transplant nephrologist/surgeon.
* No evidence of liver disease (liver enzymes < twice the upper limit of normal for each of ALT and AST, bilirubin < 2 mg/dl, albumin > 3.5 g/dl, and PT and PTT </= 1.1 x the upper limit of normal).
* Ability to comply with post-transplant regimen, including immunosuppression, insulin pump therapy and metabolic testing. Patients will be required to perform self-monitoring of blood glucose a minimum of four times daily, and provide complete records of blood glucose levels and insulin doses.
* Ability to give informed consent.
* Age greater than or equal to 18 years or less than or equal to 65 years.
* Subjects that have always been managed on a sirolimus/tacrolimus/MMF/low-dose corticosteroid (</=5mg) immunosuppressive regimen and never required conversion must provide a signed letter from their transplant nephrologist /surgeon documenting this.
* Subjects converted to a sirolimus/tacrolimus/MMF/low-dose corticosteroid immunosuppressive regimen, must provide proof of informed consent regarding immunosuppressive conversion in one of the following formats.

  * Subjects that converted to sirolimus/tacrolimus/MMF/low-dose corticosteroids (</=5mg) due to best patient care (not to qualify for islet transplantation) must provide a signed letter from their transplant nephrologists/surgeon indicating the medical reason(s) for immunosuppression conversion (with the date indicated).
  * Subjects that converted to a sirolimus/tacrolimus/MMF/low-dose corticosteroid (</=5mg) immunosuppressive regimen for the purpose of qualifying for islet transplantation must provide a signed immunosuppression conversion consent form.

Exclusion Criteria:

* Poor renal allograft function (serum creatinine > 1.6 mg/dl, creatinine clearance < 60ml/min, albumin excretion >300 mg/24hr)
* History of acute rejection related to renal graft in last 12 months or "high risk" for acute rejection (more than one previous renal transplant, PRA >25%, positive kidney crossmatch by B, T, flow cytometry)
* Current immunosuppression therapy with corticosteroids >5mg/day.
* Significant liver disease (including elevation of liver enzymes > twice the upper limit of normal for each of ALT and AST, bilirubin > 2 mg/dl, albumin < 3.5 g/dl, liver masses including portal vein thrombosis, evidence of portal hypertension, or significant, untreated gallbladder disease (i.e., gallstones).
* Significant cardiovascular disease, including non-correctable coronary artery disease with ejection fraction < 50% and/or recent myocardial infarction (within last 12 months); extensive peripheral vascular disease not correctable by surgery or untreated proliferative retinopathy.
* Recent unresolved acute infection, or chronic infection, including tuberculosis, HIV, HBV, HCV, CMV or positive skin test for TB.
* Any history of malignancy, except squamous or basal skin cancer or in situ cancer of the cervix.
* Recent history of non-compliance, or inability to demonstrate capacity to comply with strict blood glycemic control and insulin pump therapy.
* Psychiatric illness that is untreated, or likely to interfere significantly with transplantation despite treatment.
* Presence of preformed antibodies on panel reactive antibody screening > 25%.
* Body mass index (BMI) greater than 30.
* Age less than 18 years or greater than 65 years.
* Presence of a chronic disease that must be chronically treated with one or more of the following medications: glucocorticoids, diazoxide, bumetanide, haloperidol, chlorpromazine, desipramine, doxepin, imipramine, levodopa, morphine, L-asparaginase, cyclophosphamide, isoniazid, heparin, nalidixic acid, or any other agents that may adversely influence glycemic control and which may confound the interpretation of Graft Success post-transplant.
* Pregnant women, women intending future pregnancy, women of reproductive potential who are unable or unwilling to follow effective contraceptive measures for the duration of immunosuppressive therapy, and women presently breast feeding are ineligible due to the unknown effects of these drugs on the fetus and nursing infant.
* Active alcohol or substance abuse, including cigarette smoking (must be abstinent for > 3 months).
* Hyperlipidemia (total cholesterol > 260 mg/dl, LDL > 130 mg/dl, and/or triglycerides > 300 mg/dl) despite appropriate treatment.
* Anemia (Hgb < 12 g/dl) or other hematologic disorders that require medical attention.
* Increased risk of bleeding (platelet count < 80,000; INR > 1.5), other chronic hemostasis disorders, or treatment with chronic anticoagulant therapy (i.e., heparin or warfarin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Percent of subjects who have achieved insulin sufficiency post transplant. | 3, 6, 12, and 24 months

SECONDARY OUTCOMES:
Stimulated C-peptide response >0.6 ng/ml | 3, 6, 12, and 24 months
Insulin use </= 0.2 units/kg/day | 3, 6, 12, and 24 months
Reduction/elimination of hypoglycemic episodes | 3, 6, 12, and 24 months
HgAlc</= 6.5% | 3, 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fouad Kandeel, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Background] Shapiro AM, Lakey JR, Ryan EA, Korbutt GS, Toth E, Warnock GL, Kneteman NM, Rajotte RV. Islet transplantation in seven patients with type 1 diabetes mellitus using a glucocorticoid-free immunosuppressive regimen. N Engl J Med. 2000 Jul 27;343(4):230-8. doi: 10.1056/NEJM200007273430401. PMID 10911004
- [Background] Ryan EA, Paty BW, Senior PA, Bigam D, Alfadhli E, Kneteman NM, Lakey JR, Shapiro AM. Five-year follow-up after clinical islet transplantation. Diabetes. 2005 Jul;54(7):2060-9. doi: 10.2337/diabetes.54.7.2060. PMID 15983207
- [Background] Fiorina P, Folli F, Maffi P, Placidi C, Venturini M, Finzi G, Bertuzzi F, Davalli A, D'Angelo A, Socci C, Gremizzi C, Orsenigo E, La Rosa S, Ponzoni M, Cardillo M, Scalamogna M, Del Maschio A, Capella C, Di Carlo V, Secchi A. Islet transplantation improves vascular diabetic complications in patients with diabetes who underwent kidney transplantation: a comparison between kidney-pancreas and kidney-alone transplantation. Transplantation. 2003 Apr 27;75(8):1296-301. doi: 10.1097/01.TP.0000061788.32639.D9. PMID 12717219
- [Background] Fiorina P, Folli F, Zerbini G, Maffi P, Gremizzi C, Di Carlo V, Socci C, Bertuzzi F, Kashgarian M, Secchi A. Islet transplantation is associated with improvement of renal function among uremic patients with type I diabetes mellitus and kidney transplants. J Am Soc Nephrol. 2003 Aug;14(8):2150-8. doi: 10.1097/01.asn.0000077339.20759.a3. PMID 12874470